CLINICAL TRIAL: NCT04507295
Title: the Effect of Different Modes of Mechanical Ventilation on Cerebral Blood Flow During Thoracoscopic Surgeries in Neonates (RCT)
Brief Title: Cerebral Blood Flow in Neonates During Thoracoscopic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hussam Hassan, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-271-2019
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Tracheo Esophageal Fistula; Congenital Diaphragmatic Hernia
Keywords: neonates; cerebral blood flow; cerebral oximetry; VATS; VCV; PCV; ventilation
MeSH Terms: conditions — Tracheoesophageal Fistula; Hernias, Diaphragmatic, Congenital; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- volume controlled group (Active Comparator): 15 patients in is this group will be ventilated during capnothorax using volume controlled ventilation with the following parameters:
  * FIO2 of 60 %.
  * Tidal Volume (TV) of 6-8 ml/kg.
  * Respiratory rate of 30 breathes/min then the respiratory rate will be modified to maintain the ETCO2 between 30-35 mm Hg.
  * inspiratory to expiratory ratio (I: E) 1:2.
  * using a minimal Positive End Expiratory Pressure (PEEP) of 2 cm H2O.
  Interventions: Device: cerebral oximetry ( INVOS 5100 )
- pressure controlled group (Active Comparator): 15 patients in is this group will be ventilated during capnothorax using pressure controlled ventilation with the following parameters:
  * FIO2 60 %.
  * inspiratory pressure adjusted to fulfil the required TV according to the weight of the patient (6-8 ml /kg) then the insufflation pressure will be added to the driving pressure.
  * respiratory rate of 30 breathes/min then the respiratory rate will be modified to maintain the ETCO2 between 30-35 mm Hg.
  * I:E ratio of 1:1.5 .
  * Using a minimal PEEP of 2 cm H2O.
  Interventions: Device: cerebral oximetry ( INVOS 5100 )

INTERVENTIONS:
Device: cerebral oximetry ( INVOS 5100 ) — in case of critical cerebra desaturation occurred which is defined as decrease in cerebral saturation by 20% from the base line the following will be done
  1. Increase FIO2 up to 100%
  2. Increase PEEP up to 5 cmH2O
  3. Decrease insufflation pressure

SUMMARY:
the aim of this study is to compare the effect of different modes of mechanical ventilation by using volume-controlled ventilation and pressure-controlled ventilation on cerebral blood flow monitored by cerebral oximetry during thoracoscopic surgeries in neonates.

DETAILED DESCRIPTION:
The brain uses aerobic metabolism exclusively for energy production, so the brain is critically dependent on the nearly continuous delivery of oxygen to maintain cellular energy production. Normal cerebral blood flow is approximately 50 ml/100 gram of brain tissue/min. The brain represents 2% of the total body weight but it receives about 15% of the cardiac output. The brain is supplied by the circle of Willis which is formed of anastomosis between the internal carotid artery and the vertebro-basillar system. Monitoring of the CBF depends on either assessing the blood flow itself (e.g, radioactive substance and transcranial duplex) or assessing the oxygen delivery to the brain (e.g, cerebral oximetry and jugular bulb venous O2 saturation). CBF monitoring is an important parameter in both Intensive care unit and operation room in several aspects e.g, traumatic brain injury (TBI), acute stroke, carotid artery surgeries and cardiopulmonary bypass.

Cerebral oximetry is a continuous noninvasive technique that monitors the cerebral blood flow with several advantages over other CBF monitors including the ease of use and interpretation. It is painless and does not utilize ionizing radiation. The recordings provide real time information rather than single static measurements. Using the cerebral oximetry has few limitations including representing local rather than global CBF and absence of normal and cutoff values.

Thoracoscopic surgery was first introduced in 1910 and allowed a major advance in the field of thoracic surgery. Then with the improvement of the Instrumentation, thoracoscopic surgery started in the pediatric field in 1976 for simple procedures and now it is used predominantly in the pediatric thoracic surgery. The use of thoracoscope has many advantages over the open approach including using a smaller incision and reducing blood loss, postoperative pain, hospital stay and musculoskeletal deformities. Thoracoscope utilizes either one lung ventilation (OLV) or CO2 insufflation technique. In neonates the OLV technique is not suitable, so CO2 insufflation ( capnothorax ) is usually used.

Several studies were done and revealed the effect of thoracoscopy in neonate on CBF due to the effect of capnothorax which increases the intrathoracic pressure leading to decreased venous return and cardiac output, subsequently the CBF decreases, and with the increase of the insufflation pressure the decease in the CBF becomes more significant. Also the capnothorax may lead to hypercapnia which leads to changes in the CBF.

The incidence of newborn with congenital anomalies that require surgical procedure during the neonatal period is not low. With the increase of the survival rate, several studies proved that exposure of the neonates to surgery and anesthesia is associated with a higher risk of neuro-developmental delay in different aspects (sensory, motor, language, behavioral, cognitive, etc.) and thoracoscopic surgery is associated with higher risk due to the nature of the disease and the surgery. Using cerebral oximetry in addition to other routine monitors is of added value to maintain CBF within normal range to decrease the incidence of neurological injuries.

There are few studies showing that using different modes of mechanical ventilation affects CBF in neonates due to difference in several factors including effect on hemodynamics and airway pressure but there is no study comparing between volume controlled ventilation and pressure controlled ventilation. This research gap encourages us to do this study.

Preoperative assessment will be conducted on the patients the day before surgery including history taking from parents, full examination, routine laboratory investigations; in the form of CBC, coagulation profile, creatinine, urea, ALT, AST and radiological investigations; in the form of chest X-ray and echocardiography. the parents (guardians) will be consented to be included in the study & informed about the required fasting hours.

The patients enrolled in the study will be monitored all through the surgical procedure using pulse oximeter, non-invasive blood pressure and invasive blood pressure monitor (also for repeated arterial blood gases sampling), ECG, capnogram in addition to the cerebral oximetry.

Two infant probes of the cerebral oximetry will be applied to the patient on the both sides of the forehead and the monitor will display the cerebral oxygen saturation from the right and the left side of the brain digitally and in form of graph then the baseline reading of the cerebral oxygen saturation will be recorded before induction of anaesthesia.

Induction of general anaesthesia will be performed using a regimen of 1-2 µg/Kg fentanyl IV and 2-3mg/kg propofol IV then tracheal intubation is facilitated using atracurium 0.5 mg/kg IV. Ventilation will be mechanically controlled using the routine pressure-controlled mode, to maintain end tidal CO2 (ETCO2) between 30-35 mmHg.

Anaesthesia will be maintained using 1.6 % isoflurane that will be adjusted according to hemodynamics changes with top up doses of atracurium as required. After starting of gas insufflation using pressure of 4-6 mmHg and flow at 0.5 to 1.0 Liter/Minute, ventilation of patients will be modified according to the protocol of each group.

Recorded data will be analyzed using the statistical package for social sciences, version 20.0 (SPSS Inc., Chicago, Illinois, USA). Quantitative data will be expressed as mean± standard deviation (SD). Qualitative data will be expressed as frequency and percentage. The following tests will be done:

* Independent-samples t-test of significance will be used when comparing between two means.
* Mann Whitney U test: for two-group comparisons in non-parametric data.
* Chi-square (x2) test of significance will be used to compare proportions between qualitative parameters.
* The confidence interval is set to 95% and the margin of error accepted is set to 5%. So, the p-value is considered significant as the following:
* Probability (P-value) :- P-value <0.05 is considered significant. P-value <0.001 is considered as highly significant. P-value >0.05 is considered insignificant.

Sample size was calculated using G-power software. The cerebral oxygen saturation in neonates undergoing thoracoscopic surgery was derived from a previous study and was 73%±7 %.we assumed that different ventilation mode caused a difference of 10% in cerebral oxygen saturation .considering a study power of 80% and a p-value of 0.05 to be significant, the sample size was calculated to be 30 patients (15 in each group)

ELIGIBILITY:
Inclusion Criteria:

* full term neonates
* body weight more than 2500 gm

Exclusion Criteria:

* parents' refusal
* preterm neonates
* body weight less than 2500 gm
* congenital cardiac condition
* active chest condition
* congenital neurological diseases
* abnormal kidney and liver function tests

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08-08 (Estimated); Primary Completion 2020-11-08 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
cerebral saturation | during the whole duration of surgery
  the cerebral oxygen saturation ( % ) will be measured using the cerebral oximetry(INVOS 5100) and will be recorded before induction of anesthesia then every 15 minutes after induction of anesthesia and any attack of cerebral desaturation is recorded

SECONDARY OUTCOMES:
oxygen saturation ( SPO2 ) | during the whole duration of surgery
  recorded before induction of anesthesia then every 15 minutes after induction of anesthesia
arterial partial pressure of carbon dioxide ( PaCO2 ) | during the whole duration of surgery
  recorded before induction of anesthesia then every 30 minutes after induction of anesthesia
End Tidal CO2 ( ETCO2 ) | during the whole duration of surgery
  recorded after induction of anesthesia then every 15 minutes
Positive End Expiratory Pressure ( PEEP ) | during the whole duration of surgery
  any changes in PEEP in case of cerebral desaturation will be recorded
Fraction of inspired oxygen | during the whole duration of surgery
  any changes in FIO2 in case of cerebral desaturation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amel H Abo Elela, Prof, Principal Investigator — Cairo University

REFERENCES:
- [Background] Kirkness CJ. Cerebral blood flow monitoring in clinical practice. AACN Clin Issues. 2005 Oct-Dec;16(4):476-87. doi: 10.1097/00044067-200510000-00005. PMID 16269893
- [Background] Woitzik J, Dreier JP, Hecht N, Fiss I, Sandow N, Major S, Winkler M, Dahlem YA, Manville J, Diepers M, Muench E, Kasuya H, Schmiedek P, Vajkoczy P; COSBID study group. Delayed cerebral ischemia and spreading depolarization in absence of angiographic vasospasm after subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2012 Feb;32(2):203-12. doi: 10.1038/jcbfm.2011.169. Epub 2011 Dec 7. PMID 22146193
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Friedman JA, Anderson RE, Meyer FB. Techniques of intraoperative cerebral blood flow measurement. Neurosurg Focus. 2000 Nov 15;9(5):e4. doi: 10.3171/foc.2000.9.5.4. PMID 16821756
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- [Background] Kumar K, Basker S, Jeslin L, Karthikeyan C, Matthias A. Anaesthesia for pediatric video assisted thoracoscopic surgery. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):12-6. No abstract available. PMID 21804698
- [Background] Shah R, Reddy AS, Dhende NP. Video assisted thoracic surgery in children. J Minim Access Surg. 2007 Oct;3(4):161-7. doi: 10.4103/0972-9941.38910. PMID 19789677
- [Background] Dave N, Fernandes S. Anaesthetic implications of paediatric thoracoscopy. J Minim Access Surg. 2005 Mar;1(1):8-14. doi: 10.4103/0972-9941.15240. PMID 21234138
- [Background] Tytgat SH, van Herwaarden MY, Stolwijk LJ, Keunen K, Benders MJ, de Graaff JC, Milstein DM, van der Zee DC, Lemmers PM. Neonatal brain oxygenation during thoracoscopic correction of esophageal atresia. Surg Endosc. 2016 Jul;30(7):2811-7. doi: 10.1007/s00464-015-4559-1. Epub 2015 Oct 21. PMID 26490769